CLINICAL TRIAL: NCT01094925
Title: The Effectiveness of a Pre-operative Single Dose Administration of Gabapentin for Management of Post-operative Pain Following Cesarean Section: a Randomised, Double-blind, Placebo-controlled, Dose-finding Study
Brief Title: The Effectiveness of Gabapentin for Post-operative Pain Following Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Dr. Jose C.A. Carvalho, Mount Sinai Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10-01
Record Dates: First submitted 2010-03-25; First posted 2010-03-29 (Estimated); Last update posted 2011-02-23 (Estimated); Status verified 2011-02

CONDITIONS: Pain
Keywords: Cesarean section; Gabapentin
MeSH Terms: conditions — Pain | interventions — Lactose; Gabapentin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: lactose
- Gabapentin 300mg (Active Comparator)
  Interventions: Drug: Gabapentin 300mg
- Gabapentin 600mg (Active Comparator)
  Interventions: Drug: Gabapentin 600mg

INTERVENTIONS:
Drug: lactose — Single oral dose
  Arms: Placebo
Drug: Gabapentin 300mg — Single oral dose of 300mg gabapentin
  Other Names: Novo-gabapentin; Neurontin
  Arms: Gabapentin 300mg
Drug: Gabapentin 600mg — Single oral dose of 600mg gabapentin
  Other Names: Novo-gabapentin; Neurontin
  Arms: Gabapentin 600mg

SUMMARY:
Gabapentin has been very effective at treating pain after knee and hip operations, hysterectomies, and many other types of operations. A previous study at the investigators' hospital found that a single pre-operative dose of 600mg gabapentin produced a significant reduction in pain after caesarean section. However, 19% complained of sedation. The purpose of this study is to see whether a reduced dose of gabapentin will produce a similar improvement in pain scores while avoiding adverse effects such as sedation or dizziness. The objective of this study is to compare the efficacy of a single pre-operative oral dose of gabapentin 300mg, versus 600mg and placebo in women undergoing Cesarean section. The investigators' hypothesis is that gabapentin 300mg will result in decreased pain scores similar to gabapentin 600mg, but with reduced side effects.

DETAILED DESCRIPTION:
Post-operative pain is the greatest fear of women who undergo Cesarean section, and despite current analgesic regimens, this pain can be severe, impeding the mother's recovery and her ability to bond with and breastfeed her new infant. Opioids are the mainstay of treatment currently, and, although effective, these drugs have significant adverse effects, including sedation, nausea, vomiting and constipation. Non-steroidal anti-inflammatory drugs (NSAIDs) can reduce opioid consumption, but also have side effects, and are contra-indicated in a significant number of patients. Therefore there remains considerable scope to improve post-Cesarean analgesia.

It has been shown that severe acute post-operative pain after Cesarean section increases the risk of developing chronic pain and post-partum depression. A recent study showed that up to 18% of women have persistent pain after Cesarean section, and that severe acute post-operative pain is a significant risk factor.

Gabapentin is used widely to treat chronic pain, and has been demonstrated to be effective at treating acute post-operative pain following a variety of surgical procedures, with significant reductions in opioid consumption. Side effects are uncommon; the most likely are dizziness and sedation. Gabapentin does cross the placenta and into breast milk, but there is no evidence of adverse maternal or neonatal effects in women taking gabapentin during pregnancy. Gabapentin has been used successfully to treat pain in neonates.

A recent study at Mount Sinai Hospital compared a single pre-operative dose of 600mg gabapentin versus placebo in women undergoing Cesarean section. Women in the gabapentin group reported significantly improved pain scores on movement up to 48 hours after surgery. Side effects were similar in both groups apart from an increase in somnolence in the gabapentin group.

The objective of this study is to compare the efficacy of a single pre-operative oral dose of gabapentin 300mg, versus 600mg and placebo in women undergoing Cesarean section. Our hypothesis is that gabapentin 300mg will result in decreased pain scores similar to gabapentin 600mg, but with reduced side effects. We have designed a randomized, double-blind, placebo-controlled study which will aim to answer these questions. Aside from the administration of gabapentin one hour prior to surgery, there are no other changes to the standard protocol of anaesthetic care. Women will be followed up for 48 hours after surgery for assessment of pain scores and overall satisfaction. A further follow-up at three months will determine the incidence of chronic pain.

Few studies have examined the incidence of chronic pain following Cesarean section, and none have examined the impact of pre-emptive analgesia using gabapentin on the incidence of chronic pain following Cesarean section. As the rate of Cesarean section continues to increase, and there remain significant problems with current analgesic regimens, the use of gabapentin, a drug with proven effectiveness in post-surgical pain and with limited side effects, has the potential to considerably improve acute and chronic post-Cesarean pain, and lead to a widespread change in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* full term singleton pregnancy
* undergoing elective cesarean delivery

Exclusion Criteria:

* Patients unable to communicate fluently in English
* Patients with American Society of Anesthesiologists (ASA) classification of 3 or greater
* Patients with history of epilepsy or chronic pain, or of use of anti-epileptic drugs or neuropathic analgesic drugs
* Patients with a history of opioid or intravenous drug abuse
* Patients with a known allergy or contra-indication to gabapentin, or to any other drugs used in this trial
* Patients who have refused spinal anaesthesia, or those in whom it is contra-indicated
* Patients with known congenital fetal abnormalities
* Patients who have taken antacid medication in the previous 24 hours

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 126 (Actual)
Dates: Start 2010-04; Primary Completion 2010-12 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Pain score by visual analogue scale (VAS) on movement at 24 hours postoperatively | 24 hours

SECONDARY OUTCOMES:
Pain at rest and on movement by VAS, and maternal satisfaction at 6, 12, 24 & 48 hours postoperatively | 48 hours
Opioid consumption at 6, 12, 24 & 48 hours postoperatively | 48 hours
Assessment of sedation, pruritis, nausea, vomiting and dizziness on a 4-point scale (absent, mild, moderate, severe) and document treatment if required | 48 hours
Time to first maternal request for supplemental analgesia | 48 hours
Presence of pain 3 months postoperatively | 3 months
Neonatal information: Apgar scores, arterial cord blood gases, need for neonatal intensive care unit (NICU) admission | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jose CA Carvalho, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada